CLINICAL TRIAL: NCT03659487
Title: Comparison of Total and Partial Fundoplication During Surgery of Patients With Gastroesophageal Reflux Disease
Acronym: RefluxII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPN 225/01
Record Dates: First submitted 2018-08-30; First posted 2018-09-06 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Reflux, Gastroesophageal
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Intervention Model Description: Laparoscopic total (Nissen) vs posterior 270 degrees (Toupét) partial fundoplication for the treatment of gastroesophageal reflux disease.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nissen (Active Comparator): Surgery of GERD with 360 degrees total fundoplication
  Interventions: Procedure: Nissen
- Toupét (Active Comparator): Surgery of GERD with 270 degrees partial fundoplication
  Interventions: Procedure: Toupét

INTERVENTIONS:
Procedure: Nissen — Laparoscopic total (Nissen) fundoplication
  Arms: Nissen
Procedure: Toupét — Laparoscopic posterior 270 degrees partial fundoplication
  Arms: Toupét

SUMMARY:
460 patients who are scheduled for surgical treatment of gastroesophageal reflux disease (GERD) participate in the study following the usual preoperative Clinical routines (Medical history, endoscopy with biopsies, esophageal manometry with 24 hour pH (acidity) registration ). Patients are randomized to fundoplication according to Nissen or modified Toupet. Postoperatively, patients are monitored after 6 weeks 12, 36, 24 and 60 months.

DETAILED DESCRIPTION:
Patients aged 18-75 years planned for elective surgical treatment of GERD participate in the study. Patients with recurrent reflux disease following prior surgery, ASA (American Society of Anesthesiologists (ASA) Physical Status") class> 3, paraesophageal herniating and / or major herniation without reflux and those with other contraindications against laparoscopic surgery are excluded. In addition, patient completes a QOL protocol. Patients in the study are randomized to laparoscopic fundoplication performed either with a 360 degrees (Nissen) alternatively 270 degree (modified Toupét). Both of these techniques are well established clinical routines. General intubation anesthesia is standardized to all study patients. Discharge from the hospital is typically on the first postoperative day. At a visit, after 6-8 weeks for clinical control, is a QOL protocol is completed as well. After 12 and 36 months, patients undergo upper endoscopy and manometry with 24 hour pH-registration and QOL protocol completion. The latter also occurs after 24 months and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* surgery treatment for GERD
* laparoscopic surgery

Exclusion Criteria:

* previous surgery for GERD
* ASA classification >3
* paraesophageal hernias or large hiatal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2001-11 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Esophageal acid exposure | Change from baseline at 6 weeks, 12 and 36 month
  24-hour pH measurement

SECONDARY OUTCOMES:
Recurrens rates | Change from baseline at 6 weeks, 12, 36 and 60 month
  Medical journal or patients description
Dysphagia scoring | Change from baseline at 6 weeks, 12, 36 and 60 month
  Dysphagia for liquids and solids were recorded within a four-graded scale stating the frequency of dysphagia episodes with an arbitrary (empirical) cut off for clinical significance. The same dysphagia scoring was also used in a previous rct, from the same institution, comparing different types of antireflux procedures in open surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, professor, Principal Investigator — Karolinska Institut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hakanson BS, Lundell L, Bylund A, Thorell A. Comparison of Laparoscopic 270 degrees Posterior Partial Fundoplication vs Total Fundoplication for the Treatment of Gastroesophageal Reflux Disease: A Randomized Clinical Trial. JAMA Surg. 2019 Jun 1;154(6):479-486. doi: 10.1001/jamasurg.2019.0047. PMID 30840057